CLINICAL TRIAL: NCT02528123
Title: VisuMax Femtosecond Laser Small Incision Lenticule Extraction for the Correction of High Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Vision Clinic (Other)
Responsible Party: Principal Investigator, Dan Reinstein, Medical Director, London Vision Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LoVC-004
Record Dates: First submitted 2015-08-07; First posted 2015-08-19 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Myopia; Refractive Errors
Keywords: Small incision lenticule extraction (SMILE); Femtosecond laser
MeSH Terms: conditions — Myopia; Refractive Errors | interventions — Tobramycin; Dexamethasone; Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Small incision lenticule extraction (Experimental): Patients with high myopia will undergo a SMILE procedure to correct their refraction. Proxymetacaine 0.5% and Oxybuprocaine 0.4% will be used as anaesthetic during the procedure. Tobramycin and dexamethasone, and ofloxacin will be used four times a day for one week after the procedure.
  Interventions: Procedure: Small incision lenticule extraction; Drug: Tobramycin and dexamethasone; Drug: Ofloxacin; Drug: Proxymetacaine 0.5%; Drug: Oxybuprocaine 0.4%

INTERVENTIONS:
Procedure: Small incision lenticule extraction — The VisuMax femtosecond laser is used to create two interfaces that define a refractive lenticule of stromal tissue and a 2mm wide tunnel to connect the upper layer to the corneal surface. The lenticule is manually dissected and removed through the small 2mm incision without the need to create a flap as in LASIK.
  Other Names: ReLEx smile; SMILE
Drug: Tobramycin and dexamethasone — Tobramycin and dexamethasone (Tobradex) eye drops will be used four times a day for 1 week after the procedure
Drug: Ofloxacin — Ofloxacin (Exocin) eye drops will be used four times a day for 1 week after the procedure
Drug: Proxymetacaine 0.5% — Proxymetacaine 0.5% eye drops will be used as an anaesthetic during the procedure
Drug: Oxybuprocaine 0.4% — Oxybuprocaine 0.4% eye drops will be used as an anaesthetic during the procedure

SUMMARY:
The purpose of this study is to validate the safety and effectiveness of treating myopia (short-sightedness) higher than -10D using small incision lenticule extraction (SMILE) with the VisuMax femtosecond laser.

DETAILED DESCRIPTION:
Laser refractive surgery (LASIK and PRK) has been established for 25 years to treat myopia (short-sightedness). Over this time, the technology has been significantly improved to enable safe treatment of myopia up to -15D. Improvements including changing the shape of the lens of corneal tissue removed to better match the natural shape, and increasing the diameter of the applied correction to cover larger pupil sizes, have greatly reduced side-effects such as night vision glare and halos. Similarly, safety has been improved by using a laser (femtosecond laser) to create the corneal flap rather than a blade (known as a microkeratome), meaning that the cornea is reliably left with more than the safe amount of tissue.

In 2006, a new method of laser refractive surgery was introduced, small incision lenticule extraction (SMILE), which provides a minimally invasive keyhole method as it avoids the need to create a flap. In SMILE, a single laser (femtosecond laser) is used to make two curved cuts inside the cornea (without breaching the outside) that separate the lens of tissue that needs removing to focus the vision. This lens of tissue is removed in once piece (rather than evaporated as in LASIK) through a small 2mm wide tunnel to the surface.

SMILE has been used to treat short-sightedness up to -10D for more than 200,000 procedures worldwide and has been shown to achieve similar results to LASIK. However, because no flap is needed, this upper part of the cornea can also contribute strength, meaning that the cornea is stronger after SMILE than after LASIK. It is also expected that the accuracy for higher corrections using SMILE would be better than LASIK because the potential inaccuracies associated with excimer lasers (used in LASIK) are eliminated. This study will investigate the results of SMILE for myopia above -10D.

ELIGIBILITY:
Inclusion Criteria:

Only patients who are medically suitable for corneal refractive surgery can be included in the study.

* Subjects should be 21 years of age or older
* Eyes with high myopia spherical equivalent between -9.00 D up to -14.00 D, with cylinder up to 7.00 D
* The corrected distance visual acuity will be 20/40 or better in each eye pre-operatively
* Calculated sub-lenticule thickness (SLT) ≥220 µm
* Calculated total uncut stromal thickness (TUST) ≥300 µm
* Contact lens wearers must stop wearing their contact lenses at least four weeks per decade of wear before baseline measurements in case of hard contact lenses and one week before baseline measurements in case of soft contact lenses.
* Patient will be able to understand the patient information and willing to sign an informed consent
* Patient will be willing to comply with all follow-up visits and the respective examinations as specified in the flow-chart

Exclusion Criteria:

* Previous intraocular or corneal surgery of any kind on the eye being treated
* Patient not being able to lie flat in a horizontal position
* Patient not being able to tolerate local or topical anesthesia
* Autoimmune diseases
* Sicca syndrome, dry eye
* Herpes viral (herpes simplex) infections
* Herpes zoster
* Diabetes
* Pregnant or nursing women (or who are planning pregnancy during the study)
* Patients with a weight of > 135 kg
* Any residual, recurrent or acute ocular disease or abnormality of the eye, e.g.

  * Cataract
  * Suspected glaucoma or an intraocular pressure > 21 mm of Hg
  * Corneal disease
  * Corneal thinning disorder, e.g. keratoconus,
  * Pellucid marginal corneal degeneration
  * Dystrophy of the basal membrane
  * Corneal oedema
  * Exudative macular degeneration
  * Infection
* Any residual, recurrent, or active abnormality of the cornea to be treated, e.g.

  * Existing corneal implant
  * Corneal lesion
  * Unstable refraction
  * Connective tissue disease
  * Dry eye

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Z Reinstein, MD MA, Principal Investigator — London Vision Clinic
Locations (1):
- London Vision Clinic, London, United Kingdom

REFERENCES:
- [Background] Hjortdal JO, Vestergaard AH, Ivarsen A, Ragunathan S, Asp S. Predictors for the outcome of small-incision lenticule extraction for Myopia. J Refract Surg. 2012 Dec;28(12):865-71. doi: 10.3928/1081597X-20121115-01. PMID 23231737
- [Background] Reinstein DZ, Carp GI, Archer TJ, Gobbe M. Outcomes of small incision lenticule extraction (SMILE) in low myopia. J Refract Surg. 2014 Dec;30(12):812-8. doi: 10.3928/1081597X-20141113-07. PMID 25437479
- [Background] Kamiya K, Shimizu K, Igarashi A, Kobashi H. Visual and refractive outcomes of femtosecond lenticule extraction and small-incision lenticule extraction for myopia. Am J Ophthalmol. 2014 Jan;157(1):128-134.e2. doi: 10.1016/j.ajo.2013.08.011. Epub 2013 Oct 7. PMID 24112634
- [Background] Moshirfar M, McCaughey MV, Reinstein DZ, Shah R, Santiago-Caban L, Fenzl CR. Small-incision lenticule extraction. J Cataract Refract Surg. 2015 Mar;41(3):652-65. doi: 10.1016/j.jcrs.2015.02.006. PMID 25804585
- [Background] Shah R, Shah S, Sengupta S. Results of small incision lenticule extraction: All-in-one femtosecond laser refractive surgery. J Cataract Refract Surg. 2011 Jan;37(1):127-37. doi: 10.1016/j.jcrs.2010.07.033. PMID 21183108
- [Background] Ganesh S, Gupta R. Comparison of visual and refractive outcomes following femtosecond laser- assisted lasik with smile in patients with myopia or myopic astigmatism. J Refract Surg. 2014 Sep;30(9):590-6. doi: 10.3928/1081597X-20140814-02. PMID 25250415
- [Result] Sekundo W, Kunert KS, Blum M. Small incision corneal refractive surgery using the small incision lenticule extraction (SMILE) procedure for the correction of myopia and myopic astigmatism: results of a 6 month prospective study. Br J Ophthalmol. 2011 Mar;95(3):335-9. doi: 10.1136/bjo.2009.174284. Epub 2010 Jul 3. PMID 20601657

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Small Incision Lenticule Extraction
Started | 114; 187 Eyes
Completed | 113; 185 Eyes
Not Completed | 1; 2 Eyes
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 114

OUTCOME MEASURES:

1. Primary Outcome: Variability of the Refractive Predicatibility
Description: Calculate the standard deviation of the postoperative spherical equivalent, adjusted relative to the intended target, after the SMILE procedure. Analysis performed on the data from the 1 year postoperative visit. An accurate outcome is where the postoperative spherical equivalent is equal to the intended target spherical equivalent. A mean difference less than zero implies the outcome was undercorrected, whereas a mean difference greater than zero implies the outcomes was overcorrected. A smaller standard deviation represents a more accurate and more predictable outcome.
Time Frame: 1 year postop
Population: Calculate the standard deviation of the postoperative spherical equivalent, adjusted relative to the intended target, after the SMILE procedure. Analysis performed on the data from the 1 year postoperative visit. An accurate outcome is where the postoperative spherical equivalent is equal to the intended target spherical equivalent. A smaller standard deviation represents a more accurate and more predictable outcome.
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Diopters | -0.22 (0.48)

2. Secondary Outcome: Efficacy of Uncorrected Distance Visual Acuity
Description: Measure the uncorrected distance visual acuity achieved after the SMILE procedure relative to the preoperative CDVA for all eyes where the intended target refraction was emmetropia. Analysis performed on the data from the 1 year postoperative visit.
Time Frame: 1 year postop
Population: Percentage of eyes where the postop uncorrected distance visual acuity (UDVA) was within 1 line of preop corrected distance visual acuity (CDVA)
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Percentage of eyes | 87

3. Secondary Outcome: Safety of Corrected Distance Visual Acuity (Change in Corrected Distance Visual Acuity)
Description: Assess the change in corrected distance visual acuity (CDVA) before and after the SMILE procedure. Analysis performed on the data from the 1 year postoperative visit.
Time Frame: 1 year postop
Population: Percentage of eyes with loss of 2 or more lines of corrected distance visual acuity (CDVA)
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Percentage of eyes | 0

4. Secondary Outcome: Predictability of Refractive Correction
Description: Measure the postoperative refraction and calculate the deviation from the intended target in terms of spherical equivalent. Mean, standard deviation and range will be calculated. The data will also be analyzed as a scatter plot by plotting the attempted vs achieved spherical equivalent refraction. The data will also be graphically displayed as a histogram. Analysis performed on the data from the 1 year postoperative visit.
Time Frame: 1 year postop
Population: Percentage of eyes with spherical equivalent refraction within +/- 1.00 D of the intended target
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Percentage of eyes | 96

5. Secondary Outcome: Predictability of Refractive Astigmatism Correction
Description: Measure the postoperative refractive astigmatism and calculate the deviation from the intended target. Mean, standard deviation and range will be calculated. The data will also be analyzed as a scatter plot by plotting the target induced astigmatism vs the surgically induced astigmatism. The data will also be graphically displayed as a histogram. Analysis performed on the data from the 1 year postoperative visit.
Time Frame: 1 year postop
Population: Percentage of eyes with refractive cylinder up to 1.00 D after SMILE
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Percentage of eyes | 93

6. Secondary Outcome: Stability of the Spherical Equivalent Refraction
Description: Measure the postoperative refraction at 3 months and 12 months after the SMILE procedure and calculate the mean and standard deviation of spherical equivalent refraction for each time point.
Time Frame: 3 months and 1 year postop
Population: Percentage of eyes with change in SEQ more than 0.50 D between 3 and 12 months
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Percentage of eyes | 8

7. Secondary Outcome: Change in Night Vision Disturbances (Questionnaire)
Description: Provide the patient with a questionnaire to subjectively grade their quality of vision at night to assess whether this has changed after the SMILE procedure. Analysis performed on the data from the 1 year postoperative visit. A Rasch scale of 0-100 was used. A score of 0 indicates no quality of vision disturbances. A score of 100 indicates severe quality of vision disturbances. The outcome is calculated as the difference between the Rasch score before and after surgery, reported as the change in Rasch score units.
Time Frame: 1 year postop
Population: Change in total mean Rasch-scaled quality of vision score (including all symptoms) for bothersomeness
Measure: Mean (Standard Deviation); unit: scores on the Rasch scale
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
scores on the Rasch scale | 11 (23)

8. Secondary Outcome: Change in Corneal Higher Order Aberrations
Description: Measure the corneal aberrations before and after the SMILE procedure using the Atlas topographer to evaluate the change in corneal aberrations due to the surgery. Analysis performed on the data from the 1 year postoperative visit.
Time Frame: 1 year postop
Population: Change in corneal spherical aberration between 3 and 12 months
Measure: Mean (Standard Deviation); unit: Microns change spherical aberration
Units Other Than Participants: eyes
Arm/Group | Small Incision Lenticule Extraction
Number analyzed (Participants) | 113
Number analyzed (eyes) | 185
Microns change spherical aberration | 0.41 (0.16)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Small Incision Lenticule Extraction
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 10/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Incision Lenticule Extraction (N=114)
Corneal ectasia (Eye disorders) | 1 (1) — https://snomedbrowser.com/Codes/Details/14748007
Subjective visual disturbance (Eye disorders) | 9 (9) — https://snomedbrowser.com/Codes/Details/78455002

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT02528123/Prot_SAP_000.pdf